CLINICAL TRIAL: NCT00757822
Title: Prevention of Postoperative Nausea and Vomiting in Surgical Patients
Brief Title: Prevention of Postoperative Nausea and Vomiting (PONV) in Surgical Patients
Acronym: PONV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLIN-008-08S; 0167_2008I (Other Grant/Funding Number: VA)
Record Dates: First submitted 2008-09-19; First posted 2008-09-23 (Estimated); Results first posted 2016-05-13 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-04

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Dronabinol; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): dronabinol
  Interventions: Drug: Dronabinol
- Arm 2 (Active Comparator): ondansetron
  Interventions: Drug: Ondansetron

INTERVENTIONS:
Drug: Dronabinol — Dronabinol (5mg) will be administered orally (p.o.) 20-60 min pre-operatively.
  Other Names: Marinol
  Arms: Arm 1
Drug: Ondansetron — Ondansetron (4mg) will be administered intravenously (iv) intraoperatively in those patients not receiving Dronabinol.
  Other Names: Zofran
  Arms: Arm 2

SUMMARY:
This study will compare two different drug regimens (oral dronabinol versus intravenous ondanseteron) for the prevention of post-operative nausea and vomiting (PONV).

DETAILED DESCRIPTION:
Anesthesia has become remarkably safe during the past two decades, yet postoperative nausea and vomiting (PONV) continues to be a vexing problem with an unacceptably high incidence. Multiple factors including age, gender, type of surgery and anesthetic agents, perioperative opioid use and duration of anesthesia have been implicated in the cause of PONV. Several new drugs have been introduced during the last two decades to minimize PONV; however the incidence still remains significantly high, ranging from 30% during the first 24 postoperatively to 35% post discharge. Unrelenting PONV results in delayed discharge which is particularly significant after outpatient surgery. The proposed study will examine the anti-emetic properties of orally administered dronabinol given immediately prior to surgery with standard of care intravenous ondansetron given at the end of a surgical procedure in an effort to assess the need for cost effective prophylaxis of PONV.

The chemoreceptor trigger zone (CTZ) functions as emetic chemoreceptor for the vomiting centers. Many antiemetic drugs acting at the level of the CTZ are responsible for vomiting in patients receiving chemotherapy and postoperative patients. Our regimen of oral dronabinol has been proven to reduce the incidence of PONV in patients receiving chemotherapy. We intend to prove that a regimen that has been utilized in patients receiving chemotherapeutic drugs will work in patients with a high risk for developing PONV following surgery. We hypothesize that a regimen of preoperative low dose of dronabinol is superior in efficacy to a standard antiemetic in preventing the incidence of PONV, and thus will not only improve patient satisfaction but will also reduce length of stay in patients undergoing outpatient surgery.

Specific Objectives

1. Reduction of postoperative and postdischarge nausea and vomiting in ambulatory surgery patients.
2. Reduce rate of hospital admissions and length of inpatient stay after outpatient surgery.
3. Improve patient satisfaction after outpatient surgery.

Procedure After informed consent, surgical patients scheduled for outpatient abdominal surgery at the Central Arkansas Veterans Healthcare System (CAVHS) who are at high risk for developing PONV following their procedure will be randomized to receive either the study drug ( preoperative oral dronabinol-5 mg) or standard therapy ( 4 mg ondansetron intravenously at the end of surgery). The outcome measures will be the presence or absence of PONV, the severity and number of such episodes, the event count of rescue antiemetic use and patient satisfaction. All data will be recorded by personnel who are blinded to the drug regimen.

Relevance:

At CAVHS, 2/3 of our patients are scheduled for outpatient surgical procedure everyday. Our regimen will minimize postoperative and postdischarge nausea and vomiting, improve post-operative care unit (PACU) length of stay, minimize unnecessary hospital admissions, provide patient satisfaction and cost containment. The potential for application of this inexpensive intervention to other surgeries is enormous. Reducing the incidence of PONV could have a significant impact on patient satisfaction. The intervention is very low-risk, efficacious, and could substantially impact on the experience and the outcome of the Veteran undergoing surgery.

ELIGIBILITY:
Inclusion Criteria:

* The patients undergoing outpatient operations for intra-abdominal or abdominal wall procedures (e.g. hernias) under general anesthesia.
* Patients that are at increased risk for PONV based on the Koivuranta risk scoring system, with inclusion of patients having a Koivuranta risk score (K score) of 2 or more.
* Ability to give informed consent.
* Veteran eligible for treatment.

Exclusion Criteria:

* Patients <18 years old
* Patients with a history of hypersensitivity to cannabinoids or sesame oil --Patients with current substance abuse.

Substance abuse will be identified meeting one or both of the following criteria:

* a) Review the participant's medical chart to identify inpatient, residential, or outpatient treatment for alcohol or drug dependence as recorded in the Veterans Health Administration Computerized Patient Record system (CPRS) within the preceding six months.

OR

* b) Patient report. Exclude patients who report current marijuana or cocaine use within the past 30 days.

If a drug screen is clinically indicated and is positive the patient will NOT be entered into the study.

* Patients taking medications known to have significant drug-drug interactions with the prescribed drug and study drugs, Dronabinol and Ondansetron, will be reviewed in Micromedex. Micromedex is a medication database used by Central Arkansas Veterans Healthcare System (CAVHS). If the drug could have a drug-drug interaction with either dronabinol or ondansetron the patients will NOT be entered into the study. If a drug is confirmed via Micromedex not to have a drug-drug interaction, the patient will be eligible for study participation.
* Pregnant women
* Patients with prolonged QTC intervals on electrocardiogram (EKG).
* Patients enrolled in another clinical trial at the time of randomization.
* Inability to adhere to study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2009-12; Primary Completion 2013-12 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sue A Theus, PhD, Study Director — Central Arkansas Veterans Healthcare System
Locations (1):
- Central Arkansas Veterans Healthcare System-John L McClellan Memorial Veterans Hospital, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period was from 12-02-2009 to 11-20-2013. Participants were recruited during pre-surgery or preanesthesia clinic visits for elective outpatient abdominal surgery lasting at least 1 hr. Inclusion criteria included high risk for post-operative nausea and vomiting (PONV) as measured by a Koivuranta score (K score) of 2 or more.
Pre-assignment Details: 36 participants were withdrawn prior to assignment into a treatment arm: 8 participants voluntarily withdrew prior to surgery date, 2 did not meet inclusion criteria, 6 had exclusion criteria, 3 withdrawn when study was closed to enrollment, 17 were withdrawn due to cancellation or re-scheduled surgery incompatible with study schedules.
Groups:
- Arm 1: Dronabinol: dronabinol
  Dronabinol: Dronabinol (5mg) will be administered po 30-60 min prior start of surgery.
- Arm 2: Ondansetron: ondansetron
  Ondansetron: Ondansetron (4 mg) will be administered iv 20-30 min prior to end of surgery in those patients not receiving Dronabinol.
Period: Overall Study
Arm/Group | Arm 1: Dronabinol | Arm 2: Ondansetron
Started | 92 | 88
Day of Surgery (DOS) Assessment | 92 | 88
Withdrawal by Subject-no Intervention | 1 | 3
DOS Withdrawn by Investigator | 6 (No longer met inclusion criteria or developed exclusion criteria on DOS) | 11 (No longer met inclusion criteria or developed exclusion criteria on DOS)
Received Study Intervention | 85 | 74
DOS: Post-operative Assessments | 85 | 74
24-48 hr Telephone Assessment | 85 | 74
2-6 wk Post-op Assessment | 85 | 74
Data Entry, QC Assessment | 85 | 74
Withdrawn-low-risk for PONV | 12 (K score for PONV risk<2) | 9 (K score for PONV risk < 2)
Withdrawn-protocol Deviation | 9 | 8
Data Lock, Unblinding Analysis | 64 | 57
Completed | 64 | 57
Not Completed | 28 | 31

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Dronabinol: dronabinol
  Dronabinol: Dronabinol (5mg) will be administered po 20-60 min pre-operatively.
- Arm 2: Ondansetron: ondansetron
  Ondansetron: Ondansetron (4mg) will be administered iv intraoperatively in those patients not receiving Dronabinol.
- Total: Total of all reporting groups
Arm/Group | Arm 1: Dronabinol | Arm 2: Ondansetron | Total
Number analyzed (Participants) | 64 | 57 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (12.5) | 57.6 (13.2) | 57.7 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 59 | 55 | 114
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 8 | 14
  White | 58 | 48 | 106
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Risk scores for PONV [Number; unit: participants] — Post-operative Nausea and Vomiting (PONV) risk score is defined as by adding risk factors on the Koivuranta scale ( e.g. where each of the following factors: surgery lasting more than 60 minutes, female, non-smoking status, history of PONV, and history of motion sickness is assigned a value of one if present and the risk score is the summation of each factor). A K score of 0-1 represents low risk for PONV. The risk increases with K scores of 2 or more, 5 being the maximum.
  participants
    K score=2 | 44 | 35 | 79
    K score >2 | 20 | 22 | 42

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Postoperative Nausea and Vomiting
Description: The incidence of postoperative nausea (PON) and postoperative vomiting (POV) was assessed during Post-operative Care Unit (PACU) stay.
Time Frame: Post-operative Care Unit (PACU) length of stay on day of surgery (time from end of surgery to transfer to discharge unit or other hospital unit)
Population: Per protocol
Measure: Number; unit: percentage of participants
Groups:
- Arm 1:Dronabinol: dronabinol
  Dronabinol: Dronabinol (5mg) will be administered po 20-60 min pre-operatively.
- Arm 2:Ondansetron: ondansetron
  Ondansetron: Ondansetron (4mg) will be administered iv intraoperatively in those patients not receiving Dronabinol.
Arm/Group | Arm 1:Dronabinol | Arm 2:Ondansetron
Number analyzed (Participants) | 64 | 57
percentage of participants
  Incidence PACU PON | 34.4 | 29.8
  Incidence PACU POV | 12.5 | 7
Statistical Analysis 1: Comparison: Arm 1:Dronabinol vs Arm 2:Ondansetron; The incidence of PON per arm will be determined and expressed as a percentage of the total patients per arm. Treatment efficacy will be measured as the percentage-point decrease in PON in the treatment arm (Marinol) compared to the standard therapy arm (ondansetron). Null hypothesis: Marinol treatment is not superior to ondansetron treatment. We will test the statistical significance with Fisher's Exact test at a significance level of 0.05; Test type: Superiority or Other; p > 0.76, Fisher Exact; Difference in Percentages = 4.6, 90% CI 2-sided [-9.5 to 18.6]

2. Primary Outcome: Maximum Reported Post-Operative Nausea Scores on Visual Analog Scale (VAS) Scale
Description: VAS Scale: 0=no nausea, 1-3=mild nausea, 4-6= moderate nausea, 7-9= severe nausea, 10=extreme nausea usually accompanied with vomiting.
  VAS nausea score were obtained every 30 min from entry into post-operative care unit (PACU) for first 2 hrs. and then hourly until time of transfer out of PACU.
Time Frame: Post-operative Care Unit (PACU) stay from end of surgery to transfer to ambulatory unit
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: Dronabinol | Arm 2:Ondansetron
Number analyzed (Participants) | 64 | 57
percentage of participants
  No nausea (VAS score=0) | 59.4 | 70.2
  Mild Nausea (VAS score=1-3) | 15.6 | 12.3
  Moderate Nausea (VAS score =4-6) | 7.8 | 1.8
  Severe nausea (VAS score=7-9) | 7.8 | 7.0
  Extreme nausea (VAS score=10) | 9.4 | 8.8
Statistical Analysis 1: Comparison: Arm 1: Dronabinol vs Arm 2:Ondansetron; Test type: Superiority or Other; p > 0.92, Fisher Exact; One-sided Fisher's Exact test was performed comparing the percentage of subjects with at least one VAS score > 0. (Marinol>Ondansetron)

3. Primary Outcome: Post-operative Nausea and Vomiting (PONV) Incidence 24-48 Hours Post Surgery
Description: Participants were queried for presence of postoperative nausea (PON) or postoperative vomiting (POV) during the 24-48 hr window post surgery.
Time Frame: 24-48 hrs post surgery
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: Dronabinol | Arm 2:Ondansetron
Number analyzed (Participants) | 64 | 57
percentage of participants
  24-48hr PON incidence | 23.4 | 22.8
  24-48 hr POV incidence | 6.3 | 3.5
Statistical Analysis 1: Comparison: Arm 1: Dronabinol vs Arm 2:Ondansetron; Test type: Superiority or Other; p > 0.55, Fisher Exact; Difference in Percentages = 7.7, 90% CI 2-sided [-12.1 to 13.3]

4. Secondary Outcome: Post-Operative Care Unit Length of Stay (Min)
Description: Length of time in PACU (minutes) measured from end of surgery to time of transfer to ambulatory care prior to home discharge or time to hospital admission if applicable.
Time Frame: Day of surgery (time from end of surgery to transfer to ambulatory pre-discharge unit or other unit)
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Arm 1:Dronabinol | Arm 2:Ondansetron
Number analyzed (Participants) | 64 | 57
minutes | 99.5 [73 to 139] | 97.0 [70 to 150]
Statistical Analysis 1: Comparison: Arm 1:Dronabinol vs Arm 2:Ondansetron; Test type: Superiority or Other; p = 0.981, Wilcoxon Rank-Sum test

5. Secondary Outcome: Post-Surgery Hospital Admissions (All Cause) After Out-patient Abdominal Procedure
Description: Number of all-cause hospital admissions on day of elective out-patient surgery .
Time Frame: Post-operative Day of Surgery (DOS)
Measure: Number; unit: participants
Groups:
- Arm 2: Ondnasetron: ondansetron
  Ondansetron: Ondansetron (4mg) will be administered iv intraoperatively in those patients not receiving Dronabinol.
Arm/Group | Arm 1:Dronabinol | Arm 2: Ondnasetron
Number analyzed (Participants) | 64 | 57
participants
  DOS admission-observation | 3 | 3
  DOS admission- urinary retension | 4 | 3
  DOS admission-pain management | 1 | 1
  DOS admission- low SpO2 | 1 | 0
  DOS admission -intractable nausea/vomitting | 0 | 0
Statistical Analysis 1: Comparison: Arm 1:Dronabinol vs Arm 2: Ondnasetron; Test type: Superiority or Other; p > 0.90, Fisher Exact

6. Secondary Outcome: Post-operative Antiemetic Use
Description: Percentage of participants requiring post-operative anti-emetic medications.. Anti-emetic medication need was assessed during a) post-operative care unit (PACU) stay and b)during the first 48 hrs. following discharge from PACU to home or if applicable to in-patient unit.
Time Frame: End of surgery to 48 hr post surgery
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1:Dronabinol | Arm 2: Ondansetron
Number analyzed (Participants) | 64 | 57
percentage of participants
  Medication need during PACU stay | 25 | 17
  Medication need for first 48 hrs after discharge t | 3 | 4
Statistical Analysis 1: Comparison: Arm 1:Dronabinol vs Arm 2: Ondansetron; Test type: Superiority or Other; p > 0.37, Fisher Exact

7. Secondary Outcome: Patient Satisfaction: Willingness to Take Pre-operative Medication for Post-operative Nausea and/or Vomiting
Description: Percent of participants who responded that they would be willing to take preemptive medication for nausea and vomiting for subsequent surgeries when queried during post-operative follow-up interviews at 24-48 hrs or 2-6 weeks.
Time Frame: Post operative follow up interviews 24 hrs to 6 wks
Measure: Number; unit: percent of participants
Arm/Group | Arm 1:Dronabinol | Arm 2:Ondansetron
Number analyzed (Participants) | 64 | 57
percent of participants
  24-48 hr post-operative interview | 92 | 89
  2-6 week post-operative interview | 87 | 75
Statistical Analysis 1: Comparison: Arm 1:Dronabinol vs Arm 2:Ondansetron; Comparisons at 24-48 hr post-surgery. Null hypothesis: dronabinol is not superior to ondansetron in patient satisfaction; Test type: Superiority or Other; p > 0.75, FREQ Procedure
Statistical Analysis 2: Comparison: Arm 1:Dronabinol vs Arm 2:Ondansetron; Comparisons of both arms at 2-6 weeks; null hypothesis: dronabinol is not superior to ondansetron in patient satisfaction; Test type: Superiority or Other; p > 0.10, FREQ procedure

8. Secondary Outcome: Patient Satisfaction 2: Willingness to Pay Extra Money for Post-Operative Nausea and Vomiting (PONV) Preventive Medication
Description: Percent of participants willing to pay extra money for preemptive medication for PONV for subsequent surgical procedures when queried at post-operative 24-48 hr. and at 2-6 wk. follow-up interviews.
Time Frame: Post-operative follow-up interviews 24 hr to 6 weeks post surgery
Measure: Number; unit: percent of participants
Arm/Group | Arm 1:Dronabinol | Arm 2:Ondansetron
Number analyzed (Participants) | 64 | 57
percent of participants
  24-48 hr. post-op | 80 | 70
  2-6 wk post-op | 73 | 68
Statistical Analysis 1: Comparison: Arm 1:Dronabinol vs Arm 2:Ondansetron; Comparison of both group responses at 24-48 hours; Test type: Superiority or Other; p > 0.29, FREQ procedure
Statistical Analysis 2: Comparison: Arm 1:Dronabinol vs Arm 2:Ondansetron; Comparisons of both arms at 2-6 weeks; Test type: Superiority or Other; p > 0.55, FREQ Procedure

ADVERSE EVENTS:
Time Frame: 1-72 days post-surgery (e.g. 30 days post last follow-up visit at 2-6 weeks)
Description: Participant medical chart review at 2-6 weeks post operation follow-up assessment and at weekly intervals up to 30 days after last follow-up/end of participation in study.
Groups:
- Dronabinol- Experimental Therapy: Dronabinol (5mg) was administered po 30-60 min prior to start of elective abdominal surgery scheduled for same day discharge to home.
- Ondansetron-control Therapy: Ondansetron (4 mg) was administered iv 20-30 min prior to end of elective abdominal surgery scheduled for same day discharge to home.
Arm/Group | Dronabinol- Experimental Therapy | Ondansetron-control Therapy
Serious Adverse Events (participants affected / at risk) | 13/92 | 10/88
Other Adverse Events (participants affected / at risk) | 2/92 | 6/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dronabinol- Experimental Therapy (N=92) | Ondansetron-control Therapy (N=88)
overnight hospitalization secondary to unanticipated extensive surgery (Surgical and medical procedures) | 3 | 3
overnight hospitalization secondary to urinary retention (Surgical and medical procedures) | 4 | 3
overnight hospitalization secondary to excessive postoperative pain (Surgical and medical procedures) | 2 | 1
post-operative overnight hospitalization secondary to low sPO2 (Respiratory, thoracic and mediastinal disorders) | 1 | 0
post-operative complication due to surgery (Surgical and medical procedures) | 3 | 0 — Patient presented and re-hospitalized due to issues secondary to surgical procedure following discharge (e.g. infection, excessive swelling, suture rupture)
hospitalization due to co-morbid preexisting conditions (Gastrointestinal disorders) | 0 | 2 — Participant re-hospitalized within 30 days of study follow-up for further GI work-up due to pre-existing conditions.
hospitilization due to co-morbid preexisting conditions (Cardiac disorders) | 0 | 1 — iatrogenic bradycardia/hypotension
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dronabinol- Experimental Therapy (N=92) | Ondansetron-control Therapy (N=88)
Swelling at incision site (Surgical and medical procedures) | 2 (2) | 6 (6) — AE was noted if participant complained of or was seen for any swelling, redness, or other issues involving incision site and wound healing

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No